CLINICAL TRIAL: NCT01510808
Title: The Affect of Orthodontic Treatment on the Periodontal Status of Patients With Aggressive Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Tali Chackartchi, Principal Investigator, Hadassah Medical Organization
Other Study IDs: 0173-11-HMO-CTIL
Record Dates: First submitted 2012-01-11; First posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Aggressive Periodontitis
Keywords: aggressive periodontitis orthodontic stability
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Orthodontics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aggressive Periodontitis: Aggressive Periodontitis during maintenance
  Interventions: Procedure: orthodontic treatment
- aggressive periodontitis: aggressive periodontitis patients during maintenance
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: orthodontic treatment — Patients with Aggressive Periodontitis which are in the maintenance phase, had been treated for malocclusion.

SUMMARY:
Orthodontic Treatment will affect the periodontal status of periodontally treated Aggressive Periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with aggressive periodontitis in maintenance that had completed orthodontic treatment
* age 13-40
* with full records of periodontal treatment
* with full records of orthodontic treatment

Exclusion Criteria:

* smoking over 10 cigarets/day
* non controlled diabetes
* pregnancy
* alcohol consumption

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with aggressive periodontitis in maintenance that had completed orthodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-01

PRIMARY OUTCOMES:
periodontal pocket depth | one year

SECONDARY OUTCOMES:
PAR index | 1 year
  index for measuring the stability of orthodontic treatment results.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Chackartchi, DMD, Study Director — Hadassa Medical Organization - department of periodontology
Locations (1):
- Department of periodontology - Hadassah hospital, Jerusalem, Israel

REFERENCES:
- [Background] Passanezi E, Janson M, Janson G, Sant'Anna AP, de Freitas MR, Henriques JF. Interdisciplinary treatment of localized juvenile periodontitis: a new perspective to an old problem. Am J Orthod Dentofacial Orthop. 2007 Feb;131(2):268-76. doi: 10.1016/j.ajodo.2005.03.025. PMID 17276870